CLINICAL TRIAL: NCT00697801
Title: A Randomized, Double Blind, Placebo Controlled, 3 Arm, Parallel Group, Phase 2 Study Investigating the Efficacy, Tolerability and Pharmacokinetics of MAP0010 in Asthmatic Children and Adolescents Over 6 Weeks
Brief Title: Study of MAP0010 in Asthmatic Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAP0010-CL-P201
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MAP0010 low dose (Experimental): a single dose of MAP0010 low dose delivered by nebulization twice daily for 6 weeks
  Interventions: Drug: MAP0010 low dose
- MAP0010 high dose (Experimental): a single dose of MAP0010 high dose delivered by nebulization twice daily for 6 weeks
  Interventions: Drug: MAP0010 high dose
- Placebo (Placebo Comparator): Placebo delivered by nebulization twice daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MAP0010 low dose — a single dose of MAP0010 low dose delivered by nebulization twice daily for 6 weeks
  Arms: MAP0010 low dose
Drug: MAP0010 high dose — a single dose of MAP0010 high dose delivered by nebulization twice daily for 6 weeks
  Arms: MAP0010 high dose
Drug: Placebo — Placebo delivered by nebulization twice daily for 6 weeks
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy, tolerability and pharmacokinetics of 2 doses of MAP0010 (Unit Dose Budesonide) in asthmatic children/adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Male or female asthmatic children/adolescents
* 1 to 18 years of age
* FEV1 greater than or equal to 50% predicted normal (where obtainable)
* Stable but symptomatic
* Diagnosis of asthma (per NIH criteria) at least 3 months before screening OR documented exacerbation or worsening of asthma or symptoms suggestive of asthma including nocturnal asthma, within 6 months of screening OR documented SAB use more than or at least once for symptom relief during the 4 days of run in with a total symptom score greater than or equal to 1 OR greater than or equal to 1 night disturbed due to asthma symptoms in previous month.

Exclusion Criteria:

* Any other significant childhood illness.
* Participated in any investigational clinical trial within the 30 days prior to screening.
* Use of any corticosteroid within 2 weeks of screening.
* Use of oral corticosteroid within 30 days of screening or prolonged use of oral corticosteroids within 12 weeks of screening.
* Use of inhaled long acting bronchodilators.
* Presumptive or documented history of upper or lower respiratory infection within 2 weeks before screening.
* Any history of acute or severe asthma attack requiring ICU admission or ventilatory support.
* History suggestive (or diagnosis) of other concomitant lung disease.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2006-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MAP0010 High Dose | MAP0010 Low Dose | Placebo
Started | 69 | 70 | 69
Completed | 57 | 58 | 45
Not Completed | 12 | 12 | 24

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are summarized on the Intent-to-treat population (those patients with at least 1 on treatment efficacy evaluation including 1 electronic diary entry).
Groups:
- Total: Total of all reporting groups
Arm/Group | MAP0010 High Dose | MAP0010 Low Dose | Placebo | Total
Number analyzed (Participants) | 68 | 65 | 65 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (4.76) | 10.5 (4.75) | 10.2 (4.52) | 10.3 (4.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 20 | 72
  Male | 41 | 40 | 45 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daytime Composite Symptom Score
Description: The individual symptoms at each time point to be monitored are: cough, wheeze, and shortness of breath.
  The individual symptoms were scored using a four point scale:
  0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms
  Daily composite symptom score is based on the average of the individual symptom scores for a day. Daytime composite symptom score is defined as average of the last 5 days' daily composite symptom scores within the last 5 days immediately preceding the end day of that week. The range for the daytime composite symptom score is 0 (no symptoms) to 3 (severe symptoms). A negative change indicates an improvement of symptoms and a positive change indicates a worsening of symptoms.
Time Frame: baseline, week 6
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MAP0010 High Dose | MAP0010 Low Dose | Placebo
Number analyzed (Participants) | 68 | 65 | 65
units on a scale
  Baseline | 3.1 (1.90) | 2.8 (1.75) | 2.6 (1.59)
  Change from Baseline at week 6 | -0.7 (1.80) | -1.4 (1.48) | -0.6 (1.63)

2. Primary Outcome: Change From Baseline in Nighttime Composite Symptom Score
Description: The individual symptoms at each time point to be monitored are: cough, wheeze, and shortness of breath.
  The individual symptoms were scored using a four point scale:
  0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms
  Nightly composite symptom score is based on the average of the individual symptom scores for the night. Nightime composite symptom score is defined as average of the last 5 days' nightly composite symptom scores within the last 5 nights immediately preceding the end day of that week. The range for the nighttime composite symptom score is 0 (no symptoms) to 3 (severe symptoms). A negative change indicates an improvement of symptoms and a positive change indicates a worsening of symptoms.
Time Frame: baseline, week 6
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MAP0010 High Dose | MAP0010 Low Dose | Placebo
Number analyzed (Participants) | 68 | 65 | 65
units on a scale
  Baseline | 2.7 (1.96) | 2.4 (1.75) | 2.4 (1.49)
  Change from Baseline at week 6 | -0.6 (2.00) | -1.2 (1.42) | -0.4 (1.60)

3. Secondary Outcome: Change From Baseline in FEV1% Predicted
Description: The forced expiratory volume in 1 second (FEV1) is the amount forced of air exhaled in 1 second. The percent predicted is calculated for age, gender, and height. Subjects had to perform at least 3 acceptable maneuvers into a spirometer. An increase indicates an improvement (a greater volume of air expired).
Time Frame: baseline, week 6
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | MAP0010 High Dose | MAP0010 Low Dose | Placebo
Number analyzed (Participants) | 17 | 16 | 14
percentage of predicted FEV1
  Baseline | 74.8 (11.45) | 73.8 (13.10) | 65.9 (7.22)
  Change from Baseline at 6 weeks | 6.3 (9.87) | 6.3 (7.73) | 5.9 (8.73)

ADVERSE EVENTS:
Description: All patients who received any study drug and who had at least one post safety evaluation were included in the adverse event analysis.
Arm/Group | MAP0010 High Dose | MAP0010 Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/67 | 0/69
Other Adverse Events (participants affected / at risk) | 21/69 | 10/67 | 20/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MAP0010 High Dose (N=69) | MAP0010 Low Dose (N=67) | Placebo (N=69)
Nasopharyngitis (Infections and infestations) | 6 | 2 | 3
Upper Respiratory Infection (Infections and infestations) | 8 | 6 | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.